CLINICAL TRIAL: NCT06744829
Title: Prospective, Multicenter, Clinical Trial to Evaluate the Safety of the STELLA® Endogastric Balloon at 7 Months and the Balloon Introduction System
Brief Title: STELLA® Endogastric Balloon System. Evaluation of Safety and Introduction System at 7 Months.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mikromic Medical, S. L (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STELLA 2021
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Overweight/Obesity
Keywords: STELLA; Intragastric balloon; gastroscopy; Obesity; Overweight; Endoscopy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with endogastric balloon STELLA in weight loss (Experimental)
  Interventions: Device: Balloon placement and inflation and removal of the Balloon

INTERVENTIONS:
Device: Balloon placement and inflation and removal of the Balloon — STELLA Endogastric ballon will be inserted into the stomach and inflated with sterile saline solution and will remain in place for 6 months. After which the device will be removed

SUMMARY:
The main objective of the study was to evaluate the safety of the introduction of STELLA® endogastric balloon and the endogastric balloon itself at 7 months.

This investigation included screening visits and studies prior to placement, the endoscopic act of placement, the entire follow-up period while the balloon remains inside the stomach (6 months), the endoscopic act of balloon removal, as well as an additional follow-up after balloon removal of 1 month (7 months in total).

Clinical, analytical and endoscopic parameters have also been evaluated.

DETAILED DESCRIPTION:
The STELLA® endogastric balloon is a temporary, non-surgical implantable medical device designed to facilitate weight loss. It is made up of an endogastric balloon and a double-lumen probe or introducer system that allows the STELLA balloon to be placed inside the stomach. It works by partially filling the stomach, remaining freely inside, and stimulating a feeling of satiety, consequently reducing food intake.

The STELLA 2021 clinical trial was conducted in six Spanish centers and was designed as a multicentre, non-randomized, longitudinal case series clinical study to demonstrate the safety and efficacy of the STELLA® endogastric balloon.

All centers followed a common protocol. The overall aim of the study was to include a minimum of 69 patients and to collect data from these participants during the visits according to the scheduled plan.

The planned visits for this clinical investigation included baseline (comprising Screening, Baseline Visit, and Informed Consent), procedure, discharge, a telephone follow-up at 72 hours, a 10-day follow-up visit, a 3-month follow-up visit, a 6-month follow-up visit (removal of the balloon), a 7-month follow-up telephone visit, and any unscheduled visits (the investigating team could decide to conduct an unscheduled visit).

The clinical investigation included adult subjects (aged between 18 and 65 years) who were candidates for intragastric balloon placement as an aid in the treatment of their obesity. The total duration of the clinical investigation was expected to be 13 months. The end of the clinical investigation occurred when the last visit of the last enrolled subject was completed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are overweight or obese, men and women, between 18 and 65 years of age, who have failed with previous diets and who require a physical aid that increases the sensation of satiety to reduce the amount of intake and thus promote weight loss.
2. Subjects with overweight grade II (BMI between 27.00-29.99 kg/m²) and obesity grade I (BMI between 30.00-34.99 kg/m²).
3. Subjects with grade II obesity (BMI between 35.00-39.99 kg/m²) provided they do not have more than 3 major comorbidities associated with obesity.
4. Morbidly obese subjects (BMI ≥40 kg/m²) requiring weight loss by endogastric balloon prior to bariatric surgery.
5. Subjects who freely give written consent.
6. The Stella balloon is especially indicated for patients with abnormal structures of the esophagus, oropharynx or with reduced lumen size, diverticula, or other processes as long as they are benign and do not impede the passage of the endoscope.

Exclusion Criteria:

1. Patients who are participating or have participated in another clinical trial within the previous 30 days.
2. Patients who, in the opinion of the principal investigator or any of the specialists of the multicenter team, are not able to follow the instructions or to comply well with the assigned dietary treatment.
3. Systemic diseases that prevent correct monitoring.
4. Patients who do not give written informed consent to participate in the study.
5. Pregnancy and breastfeeding.
6. Patients with psychological or psychiatric disorders that, in the opinion of the psychologist, contraindicate their inclusion.
7. Unfavourable social-familial environment.
8. Patients who have previously had an endogastric balloon placed, even if it has been successful, and request the prescription of a second balloon.
9. Patients undergoing pharmacological treatment with anticoagulants, antiplatelet agents and/or NSAIDs.
10. Patients with previous surgery, bariatric or gastrointestinal surgery.
11. Previous esophageal or gastric surgery.
12. Patients with large hiatal hernia.
13. Patients with active esophagogastric pathology: Inflammatory: severe esophagitis (Los Angeles C-D), eosinophilic esophagitis, gastric and/or duodenal ulcer, Crohn's disease. Vascular: potentially bleeding lesions (varicose veins, angiomas, angiectasias). Neoplasia.
14. Anatomical alterations: digestive stenosis or occlusion.
15. Allergy to any of the implantable components.
16. Hormonal, endocrine or genetic causes of obesity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Lack of occurrence of a Severe AE related to the use of the medical device under investigation during the intervention | Patient assessment over 7 months
  Evaluate the efficacy of the STELLA® endogastric balloon on weight loss at 3 and 6 months (%TBWL, %EWL, % of patient with TBWL 10% and % of patient with EWL 25%)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Espinet Coll, MD, Principal Investigator — Digestive and Bariatric Endoscopy Unit, Hospital Universitario Dexeus
Locations (1):
- Hospital Universitario Dexeus, Barcelona, Spain

REFERENCES:
- [Derived] Espinet-Coll E, Turro-Arau R, Nebreda-Duran J, Abad-Belando R, MartinezNunez-Martinez O, Saenger F, Varas-Lorenzo M, Samaniego-Aquino FA, Diaz-Galan P, Ortega-Sabater A, Grau-Manrubia G, Lopez-Roldan G, Alberdi-Alonso JM, Galvao Neto M. Prospective, Multicenter Clinical Trial to Evaluate the Safety of the Stella(R) Intragastric Balloon at 7 Months and the Balloon Delivery System. Obes Surg. 2025 Oct;35(10):4440-4451. doi: 10.1007/s11695-025-08264-y. Epub 2025 Sep 19. PMID 40968297